CLINICAL TRIAL: NCT02803255
Title: Effect of Assist-as-needed Robot Aided Rehabilitation Strategies in Subjects With Incomplete Spinal Cord Injury
Brief Title: AAN Robotic Therapy in SCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-027F
Record Dates: First submitted 2016-05-25; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Cord Injuries
Keywords: Injuries; Spinal Cord
MeSH Terms: conditions — Spinal Cord Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Assist-As-Needed Control (Experimental): Subjects in this group will interact with a robotic exoskeleton, the MAHI Exo-II, programmed with an "adaptive mode". In this mode, the robot will continuously assist motion along pre-defined trajectories, but will employ an "assist-as-needed" protocol.
  Here, the amount of assistance provided by the robot will not be always the 100% of that required to complete the task (as in the position control mode), but only a fraction of it. The robot will continuously estimate the residual movement capabilities of the subject, depending on the specific joint addressed in the movement, and will estimate the remaining contribution needed to complete the movement following a predefined trajectory, thus avoiding to over-support motion.
  Interventions: Device: MAHI Exo-II
- Subject-Triggered Control (Active Comparator): Subjects in group B will interact with a robotic exoskeleton, the MAHI Exo-II, controlled via the subject-triggered mode, as in a previous clinical trial with the MAHI Exo II robotic system. In the subject triggered mode, the MAHIExo II is commanded to regulate joints motion following a position-control control scheme, and using as desired trajectories standardized single-joints profiles that require motion of one of the axes of the exoskeleton (i.e. elbow flexion and extension, forearm pronation and supination, wrist radial and ulnar deviation, wrist flexion and extension). The switch to position control of the exoskeleton is triggered by the application of sufficient force by the subject, in a previous phase where the robot implements a virtual wall.
  Interventions: Device: MAHI Exo-II

INTERVENTIONS:
Device: MAHI Exo-II
  Other Names: Robot-aided movement therapy

SUMMARY:
The purpose of this study is to demonstrate that a robot-aided rehabilitation protocol that follows the "assist-as needed" paradigm provide statistically significant improvements in arm and hand motor functions when compared to robot-aided protocols that passively move patients' arms along pre-defined trajectories, in patients with incomplete spinal cord injury (SCI).

ELIGIBILITY:
Twenty adults with chronic incomplete SCI (according to American Spinal Injury Association (ASIA) Impairment Scale (AIS) C-D level) will be recruited from TIRR and from the Houston area.

Inclusion Criteria:

1. Providing written informed consent prior to any study related procedures;
2. Age between 18-75 years;
3. Diagnosis of chronic complete or incomplete spinal cord injury as defined by the American Spinal Injury Association Impairment scale classification and at least for 6 months;
4. Not being involved in any specific exercise program (e.g., NMES, FES) within the previous 3 months;
5. No planned alteration in upper-extremity therapy or medication for muscle tone during the course of the study;
6. Eligibility for standard rehabilitation at the time of enrollment (i.e., absence medical comorbidities that would prevent standard rehabilitation);
7. No condition (e.g., severe arthritis, extreme shoulder pain) that would interfere with valid administration of the measures or with interpreting motor testing;

Exclusion Criteria: Subjects will be excluded if they have:

1. Any joint contracture or severe spasticity in the affected upper extremity, as measured by a Modified Ashworth Score > than 3 out of 4;
2. Subject who cannot provide self-transportation to the study location.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in ARAT score | Difference between values measured i) <1 week before treatment start and ii) <1 week after the end of the 2-4 week long treatment program

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale | Difference between values measured i) <1 week before treatment start and ii) <1 week after the end of the 2-4 week long treatment program
Change in Grip Pinch Strength Assessment | Difference between values measured i) <1 week before treatment start and ii) <1 week after the end of the 2-4 week long treatment program
Change in Graded Redefined Assessment of Strength, Sensibility and Prehension | Difference between values measured i) <1 week before treatment start and ii) <1 week after the end of the 2-4 week long treatment program
Change in Smoothness metrics | Difference between values measured i) <1 week before treatment start and ii) <1 week after the end of the 2-4 week long treatment program
  Measured via analysis of point-to-point reaching movements performed with the robot. Extracted measures include the movement-arrest-period-ratio, the spectral arc length, and the normalized average speed
Change in smoothness metrics | Difference between values measured i) treatment start day and ii) session 10 of the therapy program - 2-4 weeks after treatment start
  Measured via analysis of point-to-point reaching movements performed with the robot. Extracted measures include the movement-arrest-period-ratio, the spectral arc length, and the normalized average speed

CONTACTS AND LOCATIONS:
Overall Officials: Marcia K. O'Malley, PhD, Principal Investigator — William Marsh Rice University
Locations (2):
- United States (2):
  - Rice University, Houston, Texas
  - TIRR Memorial Hermann, Houston, Texas

REFERENCES:
- [Derived] Frullo JM, Elinger J, Pehlivan AU, Fitle K, Nedley K, Francisco GE, Sergi F, O'Malley MK. Effects of Assist-As-Needed Upper Extremity Robotic Therapy after Incomplete Spinal Cord Injury: A Parallel-Group Controlled Trial. Front Neurorobot. 2017 Jun 13;11:26. doi: 10.3389/fnbot.2017.00026. eCollection 2017. PMID 28659784